CLINICAL TRIAL: NCT01692366
Title: A Phase 2 Open-Label, Dose-Ranging Study of the Efficacy and Safety of Orally Administered SAR302503 in Japanese Patients With Intermediate-2 or High Risk Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis With Splenomegaly
Brief Title: Phase 2 Study in Japanese Patients With Intermediate-2 or High Risk Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis With Splenomegaly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD12888; U1111-1130-3710 (Other: UTN)
Record Dates: First submitted 2012-09-10; First posted 2012-09-25 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2014-09

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAR302503 300mg (Experimental): SAR302503 will be self-administered, orally, once daily, as a single agent, in consecutive, 28-day cycles at the dose level of 300mg. SAR302503 will be taken on an empty stomach at approximately the same time each day
  Interventions: Drug: SAR302503
- SAR302503 400 mg (Experimental): SAR302503 will be self-administered, orally, once daily, as a single agent, in consecutive, 28-day cycles at the dose level of 400 mg. SAR302503 will be taken on an empty stomach at approximately the same time each day
  Interventions: Drug: SAR302503
- SAR302503 500 mg (Experimental): SAR302503 will be self-administered, orally, once daily, as a single agent, in consecutive, 28-day cycles at the dose level of 500 mg. SAR302503 will be taken on an empty stomach at approximately the same time each day
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:Capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate the efficacy of daily oral doses of 300 mg, 400 mg, and 500 mg SAR302503 and combined for the response rate defined with the ≥35% reduction of spleen volume as determined by magnetic resonance imaging (MRI or computed tomography scan [CT] in patients with contraindications for MRI).

Secondary Objectives:

* To evaluate the safety of SAR302503 for both pooled (300, 400, and 500mg) and individual doses population.
* To evaluate the pharmacokinetics (PK) of SAR302503 after single and repeat-dose.
* To evaluate the effect on Myelofibrosis (MF)-associated symptoms (Key MF symptoms) as measured by the modified Myelofibrosis Symptom Assessment Form (MFSAF).
* To evaluate the durability of splenic response.
* To evaluate the effect of SAR302503 on bone marrow with regard to changes on reticulin fibrosis.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include a period to assess eligibility (screening period 28 days), followed by a treatment period of at least 1 cycle (28 days) of study treatment, and an end-of-treatment visit at least 30 days following the last administration of study drug. However, treatment may continue if patients are deriving benefit and do not have unacceptable toxicity or meet study withdrawal criteria.

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of primary or post-polycythemia vera or post-essential thrombocythemia myelofibrosis
* Myelofibrosis classified as high-risk or intermediate-risk level 2
* Enlarged spleen, palpable at least 5 cm below costal margin
* Active symptoms of myelofibrosis
* At least 20 years of age
* Eastern Collaborative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 at study entry
* Absence of active malignancy other than myelofibrosis
* Written informed consent to participate.

Exclusion criteria:

* Splenectomy.
* Any recent chemotherapy (eg, hydroxyurea), immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), immunosuppressive therapy, corticosteroids >10 mg/day prednisone or equivalent, or growth factor treatment (eg, erythropoietin), hormones (eg, androgens, danazol) within 14 days prior to initiation of study drug.
* Major surgery therapy within 28 days or radiation including spleen radiation within 6 months prior to initiation of study drug.
* Concomitant treatment with or use of pharmaceutical or herbal agents known to be moderate or severe inhibitors or inducers CYP3A4.
* Active acute infection requiring antibiotics.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
* Participation in any study of an investigational agent (drug, biologic, device) within 30 days, unless during nontreatment phase.
* Prior treatment with a JAK 2 Inhibitor.
* Treatment with aspirin in doses >150 mg/day
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
* Pregnant or lactating female. Once the lactating female stop and participate in the study, she cannot re-start feeding the baby.
* Women of childbearing potential, unless using effective contraception while on study drug. Otherwise patients must be post-menopausal (at least 1 years from last menstruation without other medical reason), or surgically sterile.
* Known active (acute or chronic) Hepatitis A, B, or C; and hepatitis B and C carriers.
* Prior history of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis, non-alcoholic steatohepatitis [NASH])

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response Rate (RR), defined as the proportion of subjects who have a ≥35% reduction as measured by MRI (or CT scan in subjects with contraindications for MRI). - Time Frame: | 24 weeks

SECONDARY OUTCOMES:
Number of patients with Serious Adverse events using NCI CTCAE v4.03, clinical parameters and vital signs | From baseline to the 30 days after last drug administration
Measurements of SAR302503 pharmacokinetic endpoints including Cmax, Tmax, and AUC0-24 | SAR302503, pre-dose and post-dose plasma collections will be obtained on Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 2, and Cycle 3 Day 1
Symptom Response Rate (SRR): Proportion of subjects with a ≥50% reduction in the total symptom score using the modified MFSAF | 24 weeks
Duration of maintenance of ≥35% reduction in spleen volume | From baseline to the 30 days after last drug administration
Percent change from baseline in spleen volume measured by MRI | 24 weeks
Percent change from baseline in spleen size measured by palpation | 24 weeks
Proportion of patients with any grade reduction in reticulin fibrosis | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Japan (7):
  - Investigational Site Number 392010, Akita
  - Investigational Site Number 392002, Bunkyō City
  - Investigational Site Number 392006, Bunkyō City
  - Investigational Site Number 392004, Sendai
  - Investigational Site Number 392008, Shinjuku-Ku
  - Investigational Site Number 392009, Shinjuku-Ku
  - Investigational Site Number 392003, Suita-Shi